CLINICAL TRIAL: NCT00447070
Title: Effect of Atazanavir on Endothelial Function in HIV-Infected Patients Compared to Standard Proteinase Inhibitors on Top of Potent Antiviral Combination Therapy
Brief Title: Effect of Atazanavir on Endothelial Function in HIV-Infected Patients
Acronym: ENDOPACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Foundation for Cardiovascular Research, Zurich (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICN 99034
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Last update posted 2009-05-27 (Estimated); Status verified 2007-03

CONDITIONS: HIV Infections; Dyslipidemia
Keywords: HIV-infection; Dyslipidemia; Endothelial Dysfunction; Atherosclerosis; Protease inhibitor; treatment experienced
MeSH Terms: conditions — HIV Infections; Dyslipidemias; Acquired Immunodeficiency Syndrome; Atherosclerosis | interventions — Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ATAZANAVIR

SUMMARY:
It is known that certain antiviral therapies, the socalled protease inhibitors, used in the treatment of HIV infection has an untowarded effect on the blood vessels, promoting early occurence of atherosclerosis. A a newer protease inhibitor, atazanavir, has been shown to have no negative effect on the levels of blood cholesterol and it is hypothesized that this may indicate that atazanavir is less prone to induce atherosclerosis. An early sign of atherosclerosis is a reduced vasomotion and this study investigate the influence of atazanavir on functionality of the conduit blood vessels compared to that of "standard" antiviral therapy.

DETAILED DESCRIPTION:
Indication: Dyslipidemia Type II in HIV-Infected Patients

Primary Objectives: Change of flow-mediated dilation in the forearm after 6 months using the protease inhibitor atazanavir in a potent antiviral therapy combination compared with a combination including current proteinase inhibitor.

Secondary Objectives: Changes in plasma lipid profiles and further clinical chemistry parameters after 6 months of treatment compared to baseline.

Study Design: This is a multicenter, observer-blind (measurements of vessel parameters and statistical evaluation), treatment-controlled, randomized, study with 2 treatment groups.

Planned Total Sample Size: (40-50) eligible randomized patients (20-25 per group) from 2-5 centers.

Subject Selection Criteria:

* Men and women, 18 to 65 years old.
* HIV-infection, documented by HIV-antibody ELISA and either positive immunoblot for HIV-antibodies or presence of HIV1 in blood.
* Two consecutive Roche Ultrasensitive Amplicor tests showing plasma HIV-1 RNA < 50 copies/ml within 60 days prior to study entry.
* CD4 count of > 100 cells/ml during 60 days prior to study entry.
* Stable antiretroviral therapy for at least 12 weeks prior to study entry (a protease inhibitor plus 2 NRTIs).
* Patient's treatment history allows, in the opinion of the investigator, atazanavir as replacement for current PI, i.e. continued viral suppression is expected based upon patient's treatment history and results of previous resistance testing, if available.
* Fasting LDL-cholesterol > 3.0 mmol/l.

Contraindications for participation:

* Known coronary artery disease, hypertension, peripheral artery disease, or cerebrovascular disease.
* Diabetes mellitus.
* Serious illness requiring systemic treatment and/or hospitalization within 14 days prior to study entry.
* Any contraindication for study medication.
* Currently on non-nucleoside reverse transcriptase inhibitors (NNRTI) (previous exposure allowed).
* Previous virologic failure on proteinase inhibitor-containing regimens which was not the consequence of poor adherence to therapy or drug adverse events; i.e. virologic failure was probably due to lack of potency of drug regimen, and may consecutively have resulted in protease resistance mutations.
* Previously documented protease resistance mutations which are known to result in cross-resistance against atazanavir.
* Any lipid lowering drugs within 4 weeks prior to study entry.
* Testosterone or anabolic steroids unless stable therapy at least 12 weeks prior to study entry.
* Systemic glucocorticoids, long-acting inhaled steroids or other immunomodulators within 30 days prior to study entry (prednisone < 10mg/day or equivalent is permitted.
* Drug or alcohol abuse, in the opinion of the investigator rendering the patient unreliable for participation.
* Participation in any other drug/treatment study.

Test Drugs:

1. Atazanavir capsules in daily standard dose (2 x 200 mg once daily) or
2. Continuation of current protease inhibitor

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 to 65 years old.
* HIV-infection, documented by HIV-antibody ELISA and either positive immunoblot for HIV-antibodies or presence of HIV1 in blood.
* Two consecutive Roche Ultrasensitive Amplicor tests showing plasma HIV-1 RNA < 50 copies/ml within 60 days prior to study entry.
* CD4 count of > 100 cells/ml during 60 days prior to study entry.
* Stable antiretroviral therapy for at least 12 weeks prior to study entry (a protease inhibitor plus 2 NRTIs).
* Patient's treatment history allows, in the opinion of the investigator, atazanavir as replacement for current PI, i.e. continued viral suppression is expected based upon patient's treatment history and results of previous resistance testing, if available.
* Fasting LDL-cholesterol > 3.0 mmol/l.

Exclusion Criteria:

* Known coronary artery disease, hypertension, peripheral artery disease, or cerebrovascular disease.
* Diabetes mellitus.
* Serious illness requiring systemic treatment and/or hospitalization within 14 days prior to study entry.
* Any contraindication for study medication.
* Currently on non-nucleoside reverse transcriptase inhibitors (NNRTI) (previous exposure allowed).
* Previous virologic failure on proteinase inhibitor-containing regimens which was not the consequence of poor adherence to therapy or drug adverse events; i.e. virologic failure was probably due to lack of potency of drug regimen, and may consecutively have resulted in protease resistance mutations.
* Previously documented protease resistance mutations which are known to result in cross-resistance against atazanavir.
* Any lipid lowering drugs within 4 weeks prior to study entry.
* Testosterone or anabolic steroids unless stable therapy at least 12 weeks prior to study entry.
* Systemic glucocorticoids, long-acting inhaled steroids or other immunomodulators within 30 days prior to study entry (prednisone < 10mg/day or equivalent is permitted.
* Drug or alcohol abuse, in the opinion of the investigator rendering the patient unreliable for participation.
* Participation in any other drug/treatment study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-08; Study Completion 2006-05

PRIMARY OUTCOMES:
Change of flow-mediated dilation in the forearm after 6 months using the protease inhibitor atazanavir in a potent antiviral therapy combination compared with a combination including current proteinase inhibitor.

SECONDARY OUTCOMES:
Changes in plasma lipid profiles and further clinical chemistry parameters after 6 months of treatment compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Weber, Prof., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Infectiology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Result] Flammer AJ, Vo NT, Ledergerber B, Hermann F, Gamperli A, Huttner A, Evison J, Baumgartner I, Cavassini M, Hayoz D, Quitzau K, Hersberger M, Sudano I, Ruschitzka F, Luscher TF, Noll G, Weber R. Effect of atazanavir versus other protease inhibitor-containing antiretroviral therapy on endothelial function in HIV-infected persons: randomised controlled trial. Heart. 2009 Mar;95(5):385-90. doi: 10.1136/hrt.2007.137646. Epub 2008 Jul 24. PMID 18653575